CLINICAL TRIAL: NCT05982470
Title: Effect of Menopause Hormone Therapy In Postmenopausal Women With CeRebral Small Vessel DiseAse And Mild Cognitive DecLinE
Brief Title: Effect of Menopause Hormone Therapy In Postmenopausal Women With CSVD And MCI
Acronym: MIRACLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2023-117
Record Dates: First submitted 2023-07-18; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Small Vessel Diseases; Postmenopausal Symptoms; Mild Cognitive Impairment; White Matter Hyperintensity
Keywords: cerebral small vessel diseases; Menopausal Hormone Therapy; Postmenopausal Symptoms; Mild Cognitive Impairment; White Matter Hyperintensity
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): Estradiol gel 2.5 g (containing 17β estradiol 1.5mg) once daily (percutaneous application)* in combination with progesterone soft capsules 100mg once daily (oral) for 12 months
  Note :
  * Usage and dosage of estradiol gel: A dose of ruler is applied to the skin of the arm, shoulder, head and neck, abdomen, thigh or face every morning or evening. It is dry about two minutes after application. It is non-irritating, colorless, or milky white and tasteless, and is best used after bathing.
  Interventions: Drug: Estradiol Gel; Drug: Progesterone Soft Capsule
- control group (Placebo Comparator): Estradiol placebo gel 2.5g (containing 17β estradiol 0mg) once daily (percutaneous application) *in combination with progesterone placebo soft capsules(containing progesterone 0mg) 100mg once daily (oral) for 12 months
  Note :
  * Usage and dosage of estradiol placebo gel : A dose of ruler is applied to the skin of the arm, shoulder, head and neck, abdomen, thigh or face every morning or evening. It is dry about two minutes after application. It is non-irritating, colorless, or milky white and tasteless, and is best used after bathing.
  Interventions: Drug: Estradiol Placebo Gel; Drug: Progesterone Placebo Soft Capsule

INTERVENTIONS:
Drug: Estradiol Gel — Estradiol gel 2.5 g (containing 17β estradiol 1.5mg) once daily (percutaneous application) for 12 months
  Arms: treatment group
Drug: Estradiol Placebo Gel — Estradiol placebo gel 2.5 g (containing 17β estradiol 1.5mg) once daily (percutaneous application) for 12 months
  Arms: control group
Drug: Progesterone Soft Capsule — Progesterone soft capsules 100mg once daily (oral) for 12 months
  Arms: treatment group
Drug: Progesterone Placebo Soft Capsule — Progesterone placebo soft capsules 100mg once daily (oral) for 12 months
  Arms: control group

SUMMARY:
The objective of this clinical trial is to explore the efficacy of menopausal hormone therapy in early menopausal women with CSVD and MCI.

The main questions it aims to answer are:

* The efficacy of menopausal hormone mainly estrogen therapy for early menopausal women with CSVD and MCI
* The role of MHT in delaying the progression of cognitive function, CSVD imaging features, and other clinical symptoms and the potential pathophysiological mechanisms.

Participants will be divided randomly into two groups taking MHT drugs and placebo respectively and followed up for 12 months to collect relevant clinical data.

DETAILED DESCRIPTION:
Cerebral small vessel disease (CSVD) is a common chronic whole brain syndrome in middle-aged and elderly people, mainly involving small-arteries, arterioles, capillaries, venules and small-veins in the brain. CSVD mainly relies on typical imaging features for diagnosis. Aging is the most common risk factor for CSVD. With the acceleration of China's aging process, the Disease burden of CSVD is increasing.

Menopause refers to the permanent cessation of menstruation caused by ovarian failure. During menopause, drastic changes in hormones can have a series of effects on women.Research shows that menopause is an independent risk factor for WMH. Meanwhile, menopause is significantly associated with cognitive impairment, especially with decreased learning, memory, and attention. Menopause can also cause changes in cerebral hemodynamics, damage to the integrity of the Blood-brain barrier and atrophy of cortical structures.

Estrogen not only plays a crucial role in maintaining vascular function, but also has significant neuro-protective effects. Estrogen-based menopausal hormone therapy (MHT) is essentially a treatment measure taken to compensate for ovarian failure caused by aging.

However, it is still unclear whether MHT can effectively alleviate CSVD symptoms and delay CSVD progression. The MHT treatment plan may also be an important reason for the inconsistent conclusions on the impact of MHT on cognitive function in various clinical studies. In previous clinical studies, the MHT regimen was oral estrogen (with or without Progestogen).

Based on the above research background, MHT, especially the MHT regimen using transdermal estrogen, may be an effective treatment method to improve and alleviate the rapid progression of CSVD in perimenopausal women(without contraindications). So far, there have been no RCT studies evaluating the effectiveness and safety of MHT in CSVD patients internationally. Therefore, more research is needed to provide stronger evidence and provide new directions and basis for the treatment of CSVD.

Participates who met the inclusion criteria were randomly divided into two groups. Participants were treated with MHT/placebo followed up for 12 months, and collected and analyzed relevant clinical data to evaluate the efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. 40 ≤ age < 60 years
2. Female;
3. 1 year ≤ Natural menopause≤ 6 years;
4. FSH ≥ 35 miu/ml and E2 ≤ 25 pg/ml;
5. Head MRI shows CSVD-related image changes, meet one of the following:

   1. Parventricular or deep brain white matter hyperintense, Fazekas ≥ 2；
   2. Parventricular or deep brain white matter hyperintense, Fazekas = 1, with more than 2 vascular risk factors (hypertension, hyperlipidemia, type 2 diabetes, obesity, current smoking);
   3. Parventricular or deep brain white matter hyperintense, Fazekas = 1, with more than 1 vascular-derived lacunae;
   4. Recent small subcortical infarction within the last 3 months
6. Mild cognitive dysfunction (18 ≤ MoCA <26);
7. Independent in daily life (mRS ≤ 1）
8. Sign informed consent.

Note:

1. Natural menopause: The self-reported last menstrual date of the subject
2. CSVD related image changes: evaluated according to the STRIVE2 standard issued in 2023;
3. Fazekas score: The total score is 6 , which is the sum of Fazekas scores for subcortical and periventricular white matter lesions;
4. Recent subcortical small infarcts: lesions with a diameter of<20mm in the subcortical, basal ganglia, or brainstem regions that exhibit high signal intensity (ADC diffusion limitation) on DWI imaging, with or without corresponding clinical symptoms; With new clinical symptoms, FLAIR hyperintense lesions (<20mm in diameter) in subcortical, basal ganglia or corresponding parts of pons can be seen in FLAIR sequence of head MRI.
5. MoCA: Montreal Cognitive Assessment; If the subject's education period ≤ 12 years, then increase by 1 point, with a maximum score of 30 points;
6. mRS: Modified Rankin Scale

Exclusion Criteria:

1. Inheritable CSVD, such as CADASIL, CARASIL, etc.
2. Confirmed neurodegenerative diseases, such as AD and PD;
3. Clear non-vascular white matter lesions, such as multiple sclerosis, adult brain white matter dysplasia, metabolic encephalopathy, etc.
4. History of intracranial hemorrhagic disease within the recent 6 months, including cerebral parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural / extradural hematoma, etc., as well as untreated aneurysms (diameter> 3mm) and cerebrovascular malformations.
5. Cardiovascular and cerebrovascular events within the past 6 months, such as myocardial infarction, unstable angina pectoris, cerebral infarction, etc.
6. Previously received or initiated menopausal hormone therapy.
7. Previous Hysterectomy
8. Vaginal bleeding of unknown origin
9. Intra- and extra- cranial Atherosclerosis large artery stenosis (50-99%) or occlusion.
10. Active venous or arterial thromboembolic diseases, such as Deep vein thrombosis, Pulmonary embolism, myocardial infarction, angina pectoris or congestive heart failure, in the last 6 months.
11. Used drugs and Phytoestrogen supplements that affect estrogen levels in the past 3 months, such as soybean concentrate or extract, Kuntai capsule, Dingkundan, Lifumin, etc.
12. Endometrial hyperplasia, vaginal ultrasound indicates endometrial ≥ 5mm (note: those confirmed as benign lesions by pathology can be included).
13. Severe liver and kidney dysfunction: severe liver dysfunction refers to Alanine transaminase>3 times the upper limit of normal value or cereal grass Transaminase>3 times the upper limit of normal value; Severe renal insufficiency refers to blood creatinine>3.0 mg/dl (265.2 μmol/L) or glomerular filtration rate<30 ml/min/1.73m^2;
14. Hypertension is still difficult to control after standardized treatment (blood pressure>160/100mmHg); Type 2 diabetes is still difficult to control after standard treatment (Glycated hemoglobin ≥ 8%).
15. Known or suspected to have sex hormone dependent malignant tumors, such as breast cancer, endometrial cancer, cervical adenocarcinoma, ovarian cancer, and meningioma.
16. Suffering from severe organic diseases with an expected survival time of<5 years.
17. Other situations that are not suitable for menopausal hormone treatment, such as porphyria, otosclerosis, etc.
18. Mental disorders diagnosed according to DSM-5 diagnostic criteria, or previous mental system diseases that cannot be fully communicated.
19. Allergies to the active ingredients or any of the excipients of the research drug.
20. Contraindications to MRI examination, such as Claustrophobia, metal implants in the body, etc.
21. Unable to cooperate in completing follow-up due to geographical or other reasons.
22. Situations deemed unsuitable by other researchers to participate in the study.
23. Participating in other interventional clinical trials. -

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Early menopause of female
Enrollment: 328 (Estimated)
Dates: Start 2023-08-18 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
the changes in the Montreal Cognitive Assessment (MoCA; range, 0-30; with lower scores indicating more severe cognitive impairment) scores 1 year after randomization compared to baseline | 1 year after randomization
  the changes of the Montreal Cognitive Assessment (MoCA; range, 0-30; with lower scores indicating more severe cognitive impairment) scores

SECONDARY OUTCOMES:
the changes in each cognitive domain estimated bythe Montreal Cognitive Assessment (MoCA; range, 0-30; with lower scores indicating more severe cognitive impairment) sub-items 1 year after randomization compared to baseline | 1 year after randomization
  the changes in each cognitive domain estimated by the Montreal Cognitive Assessment (MoCA; range, 0-30; with lower scores indicating more severe cognitive impairment) sub-items
the changes of modified Kupperman scores (0-63; with higher scores indicating more severe symptoms) 1 year after randomization compared to baseline | 1 year after randomization
  the changes of modified Kupperman scores (0-63; with higher scores indicating more severe symptoms)
the changes of Pittsburgh sleep quality index(PSQI; with higher scores indicating more severe sleep quality) 1 year after randomization compared to baseline | 1 year after randomization
  the changes of Pittsburgh sleep quality index(PSQI; with higher scores indicating more severe sleep quality)
the changes of Hamilton Depression Scale(HAMD; ranges, 0-54; with higher scores indicating more severe depression) 1 year after randomization compared to baseline | 1 year after randomization
  the changes of Hamilton Depression Scale(HAMD; ranges, 0-54; with higher scores indicating more severe depression)
the changes of Hamilton Anxiety Scale(HAMA; ranges, 0-56; with higher scores indicating more severe anxiety) 1 year after randomization compared to baseline | 1 year after randomization
  the changes of Hamilton Anxiety Scale(HAMA; ranges, 0-56; with higher scores indicating more severe anxiety)
the changes of the volume of white matter hyperintensity 1 year after randomization compared to baseline | 1 year after randomization
  the changes of the volume of white matter hyperintensity
Serum levels of estradiol 1 year after randomization compared to baseline | 1 year after randomization
  Serum levels of estradiol
Serum levels of follicle stimulating hormone 1 year after randomization compared to baseline | 1 year after randomization
  Serum levels of follicle stimulating hormone

OTHER OUTCOMES:
the incidence of combined outcome (including recent small subcortical infarct and combined vascular events) 1 year after randomization | 1 year after randomization
  the incidence of combined outcome (including recent small subcortical infarct and combined vascular events)

CONTACTS AND LOCATIONS:
Overall Officials: yilong wang, MD,PhD, Principal Investigator — Beiiing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China